CLINICAL TRIAL: NCT05663814
Title: Factors Affecting Prognosis of Open Globe Injuries in Assiut University Hospitals
Brief Title: Factors Affecting Prognosis of Open Globe Injuries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Natag Riad, principal investigator, Assiut University
Other Study IDs: Open globe injuries
Record Dates: First submitted 2022-11-19; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Open Globe Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
: Detailed history should be taken from the patients ( age ,sex ,location of accident (rural or civil) , time of injury , mode of trauma, exact mechanism of injury ) Examination at baseline to determine location and extent of injury. Associated injuries e.g. cataract ,hyphema . Assessment for other life threatening injuries. Exclusion of IOFB. The presenting visual acuity should be recorded in injuried and uninjuried eye. Fundus examination if possible. The pupils should be examined for RAPD (in blunt trauma searching post traumatic optic neuropathy) Slit lamp examination at presentation to detect extent of damage. {type of wound ( corneal ,scleral ,or corneoscleral ) , prolapsed uveal tissue presence of hyphema ,sublaxated or dislocated lens ,prolapsed vitreous } Investigations done before repair (e.g. CT orbit ) Time of primary repair should be recorded. Follow up visits at 1 day, 1 week, 1 month, 3 months for :-

1. For healing.
2. Suture status.
3. Detailed slit lamp and fundus examination.
4. UCVA
5. BCVA
6. Investigations including:- B scan if hazy media OCT if clear media
7. Refraction if possible Post operative complications and 2ry interventions

Aim of study :

predict the final visual outcome of open globe injuries. Assess most common modes of trauma in open globe injuries. Assess postoperative complications and secondary intervention

DETAILED DESCRIPTION:
Open globe injury (OGI) is defined as a full-thickness wound of the eyewall. Its global incidence rate is 3.5 per 100,000 persons per year , but the rates vary between countries and populations depending on the socio-economic status, education, and lifestyle. These injuries result in poor visual outcome and cause severe ocular morbidity and blindness. Unexpected and sudden occurrence of the injury may cause a psychosocial problem, permanent changes in quality of life, career and plans of the sufferers. These problems also affect not only the patients, but also all their family members.

Despite the improvement in instrumentation and ocular surgery techniques, and increased awareness of occupational safety, OGI patients still exhibit poor visual prognosis. And sometimes, they can not perceive the seriousness of the injury. Therefore, the estimation of visual prognosis is very beneficial in managing the expectation of patients and establishing a treatment strategy. Many factors, such as the type of injury, mechanism of injury, the location of the wound, and posterior segment involvement, have been suggested to influence the visual prognosis in OGI.

Ocular penetrating and perforating injuries (commonly referred to as open globe injuries) can result in severe vision loss or loss of the eye. Penetrating injuries by definition penetrate into the eye but not through and through--there is no exit wound. Perforating injuries have both entrance and exit wounds. Typically, to constitute one of these injuries, a full-thickness rupture of the cornea and/or sclera must be present. Open globe rupture, in contrast, refers to blunt injury of the eye causing globe collapse. This typically occurs at the limbus and near the equator behind the recti muscles insertions, where the sclera is thinnest.

ELIGIBILITY:
Inclusion Criteria:

1. Age + 6
2. Laceration, incised injury ,Penetrating and perforating injuries
3. Rupture globe

Exclusion Criteria:

1. age less than 6
2. patients unwilling to participate in study
3. patients with disorganized globes

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any patient more than 6 years presented with open globe injury
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Factors affecting prognosis of open globe injuries in Assiut university hospitals | 1 year
  Final visual acuity in Snellen chart

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Soliman, Prof, Principal Investigator — Assiut University

REFERENCES:
- [Background] Zhou Y, Chang P, Abdelmalik B, Mayer Z, Shah A, Steigleman WA. Prognosis of Open Globe Injuries at a Tertiary Referral Center: The Modified Florida Ocular Trauma Score. Am J Ophthalmol. 2022 Dec;244:152-165. doi: 10.1016/j.ajo.2022.08.015. Epub 2022 Aug 23. PMID 36007553